CLINICAL TRIAL: NCT02335190
Title: Ultrasound-guided Sacroiliac Joint Radiofrequency Ablation: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: University of Toronto (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Eldon Loh, Assistant Professor, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8368-US
Record Dates: First submitted 2015-01-05; First posted 2015-01-09 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Sprain of Sacroiliac Ligament; Low Back Pain; Osteoarthritis Nos, of Sacroiliac Joint
Keywords: Sacroiliac joint; Radiofrequency ablation; Ultrasound
MeSH Terms: conditions — Low Back Pain; Joint Diseases | interventions — Radiofrequency Ablation; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PSN block and RF ablation (Experimental): Participants will first undergo a lidocaine block of the PSN at the lateral crest under ultrasound guidance. On a separate visit, participants will then undergo ablation of the PSN at the lateral crest under ultrasound-guidance.
  Interventions: Procedure: Radiofrequency ablation; Procedure: Sensory block; Drug: Lidocaine

INTERVENTIONS:
Procedure: Radiofrequency ablation — RF ablation will be performed using 2 Nimbus multitined electrodes in a bipolar configuration. The electrodes will be placed along the lateral crest using a leap-frogging technique from the inferomedial aspect of the PSIS to the third transverse sacral tubercle at 1.5-2 cm intervals at the skin surface. A radiofrequency current will be passed for 120 seconds per site resulting in thermal coagulation of the plexus. Prior to performing the thermal lesion, electrical stimulation at 2 Hz and 2.0 V will be administered.
  Other Names: RF ablation
Procedure: Sensory block — Participants will undergo a lidocaine block of the PSN at the lateral crest under ultrasound guidance. 0.5 mL of 2% lidocaine will be injected from the inferomedial border of the PSIS to the third transverse sacral tubercle at approximately 1.5 cm intervals along the skin surface.
  Other Names: Posterior sacral network block; PSN block
Drug: Lidocaine

SUMMARY:
The sacroiliac (SI) joint is a common source of low back pain. Radiofrequency ablation (RFA) can be used to treat low back pain from the SI joint , and is often recommended by physicians to provide long lasting pain relief. However, the use of RFA for SI joint pain has not been as successful as RFA for pain in other areas of the back and neck. X-ray guidance (fluoroscopy) is currently used to perform this procedure. Under fluoroscopy, however, it can be difficult for physicians to identify necessary landmarks, and there are risks to the patient because of radiation exposure. In contrast, ultrasound may provide better image guidance than fluoroscopy, and there is no radiation risk. The purpose of this study is to examine if ultrasound guided SI joint RFA is effective.

DETAILED DESCRIPTION:
Background:

This study will examine the effectiveness of sacroiliac joint (SIJ) diagnostic sensory blocks and radiofrequency ablation (RFA) under ultrasound guidance. The sacroiliac joint (SIJ) is estimated to be the source of pain in 10-27% of patients suffering from mechanical low back pain. When pain is refractory to conventional treatments (such as activity modification, exercise, physical therapy, chiropractic, anti-inflammatory and analgesic medications and corticosteroid injections), radiofrequency ablation (RFA) is a treatment option in carefully selected individuals.

Current practice is to perform the SIJ posterior sensory blocks and RFA under fluoroscopic guidance. Research has confirmed that SIJ RFA can provide significant relief, however, the success rate and magnitude of relief are variable. Part of this variability may relate to the challenging nature of identifying key anatomical landmarks under fluoroscopy - their location may not be clearly evident with fluoroscopy particularly if the patient is obese, has low bone mineral density or has abundant bowel gas and/or stool in the pelvis.

A recent cadaveric study by our research group has clarified the sensory innervation of the SIJ and the findings have implications for currently practiced SIJ sensory block and RFA procedures. The study confirmed that the posterior sacral network innervates the SIJ and runs along the lateral crest of the sacrum between the S1 and the S3 lateral sacral tubercles. Inasmuch as the lateral sacral crest is predictably and clearly visible on ultrasound, posterior sacral network (PSN) SIJ sensory blocks and RFA under ultrasound guidance may be feasible using the lateral sacral crest as the key anatomical structure.

No clinical studies have been done that use ultrasound guidance for SIJ RFA. There are numerous advantages to ultrasound-guided SIJ sensory block and RFA. Significantly, patients would no longer be exposed to ionizing radiation for their SIJ procedures. With an improved understanding of SIJ sensory innevation and technical improvements in RFA electrodes, we hypothesize that ultrasound guided SIJ diagnostic sensory blocks and RFA will lead to clinically significant outcomes that will be at least comparable to conventional fluoroscopic-guided techniques.

Objectives:

1. To evaluate the relative effectiveness of ultrasound-guided PSN sacroiliac joint sensory block compared to fluoroscopic-guided lateral branch sacroiliac joint block.
2. To evaluate the relative effectiveness of ultrasound-guided PSN sacroiliac joint radiofrequency ablation compared to fluoroscopic-guided lateral branch sacroiliac joint RFA.

Methodology:

This study is a prospective cohort study examining the effectiveness of ultrasound-guided SIJ sensory block and RFA of the PSN, compared to fluoroscopic guided SIJ RFA. Participants will first undergo a local anesthetic block under ultrasound guidance to determine the predictive value of this test for SIJ RFA; they will then undergo the SIJ RFA procedure. For some patients in this study, this will be a repeat RFA procedure as they would have had a previous fluoroscopic-guided SIJ RFA with success, but subsequent return of their pain.

SIJ Sensory Block: Eligible study subjects will initially undergo a lidocaine block of the PSN at the lateral crest under ultrasound guidance. Their index pain intensity prior to the block must be >2/10. Under ultrasound guidance, 0.5 mL of 2% lidocaine will be injected from the inferomedial border of the PSIS to the third transverse sacral tubercle at approximately 1.5 cm intervals along the skin surface. Following the local anesthetic block, the subject will be asked to complete a pain diary for 6 hours. Specifically, their baseline pain will be reassessed and their ability to perform functional activities will also be assessed over that time period. The results of this block will be compared to the results of conventional blocks done under fluoroscopy.

SIJ RFA: Ultrasound-guided RFA of the PSN will be performed using the same technique as the local anesthetic block with the exception that 2 Nimbus multitined electrodes will be used in a bipolar configuration. The electrodes will be placed along the lateral crest using a sequential, leap-frogging technique from the inferomedial aspect of the PSIS (at or just above the level of the S1 dorsal sacral foramen if visible, or the S1 spinous process if not) to the third transverse sacral tubercle at 1.5-2 cm intervals at the skin surface. A radiofrequency current will be passed for 120 seconds per site thus raising the temperature at the dorsal periosteum and adjacent soft tissue to 80°C resulting in thermal coagulation of the plexus. Prior to performing the thermal lesion, electrical stimulation at 2 Hz and 2.0 V will be administered. If the patient perceives, or the operator observes muscle contraction of the leg or anal sphincter, no radiofrequency current will be applied and the needle tip will be adjusted to a position away from where the sacral nerve roots may lie.

Analysis:

The effectiveness of ultrasound-guided sensory blocks and RFA will be directly compared to the effectiveness of fluoroscopic-guided sensory blocks and RFA. In patients who have had the SIJ RFA procedure previously, their current ultrasound-guided PDQQ-S scores will be compared to their previous fluoroscopic-guided PDQQ-S results. In patients who are receiving the SIJ RFA procedure for the first time, a database of SIJ RFA PDQQ-S scores of patients treated over the past 5 years with the fluoroscopic-guided RFA technique is available for comparison. Their results will be compared to age and pre-RFA matched patients from the database.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Clinical presentation compatible with SI joint origin pain (back pain below L5; localized to the SI joint area; >2 positive of 5 SI joint provocative tests).
* >50% index pain relief with at least one SIJ intra-articular local anesthetic block and at least one SIJ lateral branch block using the conventional fluoroscopically guided lateral branch block technique. Pain diary records for these interventions need to be on file.

Exclusion Criteria:

* Under 18 years of age
* Presence of clinical and investigative evidence of inflammatory spondyloarthropathy, fibromyalgia, radiculopathy, symptomatic spinal stenosis, facetogenic or discogenic low back pain, generalized infection, localized infection in the area of the low back/SIJs, coagulopathy or anticoagulation, allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale for pain | Hourly for 6 hours post-block
  Pain diary scores for first 6 hours post-block
Pain Disability Quality-of-Life Questionnaire (PDQQ-S) | 2 months post-RF procedure
  The PDQQ-S is a 6 item questionnaire exploring 3 domains: pain, disability and quality-of-life. There are 2 questions for each domain and each is graded from 0 to 10 using a numerical rating scale. Ultrasound-guided SIJ RFA results will be compared to previous fluoroscopic-guided SIJ RFA results at 2 months.

SECONDARY OUTCOMES:
Pain Disability Quality-of-Life Questionnaire (PDQQ-S) | 6, 9, 12, 16, 20 and 24 months post-RF procedure
  Secondary outcome will be the duration of improvement on the PDQQ-S, and will be measured by repeat administration of the PDQQ-S every 3-4 months up to 24 months post-procedure. If there is ongoing, clinically significant relief at 6 months (>30% improvement in pain intensity and/or at least 2 point improvement on the pain severity question (question #1) of the PDQQ-S), patients will be reached by phone to complete the PDQQ-S at 3-month intervals up to 12 months post-RFA and then at 4-month intervals up to 24 months, or until their pain intensity returns to baseline (<30% improvement and/or <2 point improvement on question 1 of the PDQQ-S on 2 consecutive follow-ups), whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Eldon Loh, MD, Principal Investigator — Western University; Robert S Burnham, MD, M.Sc., Principal Investigator — University of Alberta
Locations (1):
- St. Joseph's Pain Clinic, London, Ontario, Canada